CLINICAL TRIAL: NCT06185790
Title: The Effect of a Low Carbohydrate- High Fat Diet on Clinical Symptoms and Gut Microbiome in m.3243A>G Related Mitochondrial Diabetes
Brief Title: MItochondrial Diabetes LOw Carb- Diet Study
Acronym: MIDLOC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Collaborators: Stichting Stofwisselkracht (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: NL85039.091.23
Record Dates: First submitted 2023-11-30; First posted 2023-12-29 (Actual); Last update posted 2025-01-13 (Actual); Status verified 2024-12

CONDITIONS: Mitochondrial Diseases; Diabetes-Deafness Syndrome Maternally Transmitted
Keywords: low carbohydrate high fat diet; gut microbiome; mitochondrial diabetes
MeSH Terms: conditions — Mitochondrial Diseases; Noninsulin-dependent diabetes mellitus with deafness

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- LCHF diet (Experimental): Participants will adhere to a low-carb high-fat diet for 12 weeks,defined by a carbohydrate intake of 50-100 grams per day.
  Interventions: Other: LCHF diet
- Control (No Intervention): Participants will follow their usual diet for 12 weeks.

INTERVENTIONS:
Other: LCHF diet — Low-carb high-fat (LCHF) diet
  Arms: LCHF diet

SUMMARY:
In daily practice, doctors and dietitians in the clinic receive many questions in general from patients with a Mitochondrial Disease (MD), and more specific whether nutritional changes can alleviate their symptoms. Mitochondrial Inherited Diabetes and Deafness (MIDD) is due to a mitochondrial mutation at the m.3243A>G locus. Nutrition is known to affect disease burden in MIDD. Which diet does this best is unknown. Very low carbohydrate high fat diets improve mitochondrial function in isolated cells and in mice. Whether it does so in people with MIDD is unknown. Therefore, the objective of the study is to explore the effect of a low carbohydrate- high fat diet (LCHF) on clinical symptoms (Goal Attainment Scaling) and gut microbiome in patients with MIDD due to the m.3243A>G mutation. A total of 20 adult patients with the above mentioned characteristics will be randomized to receive first usual care during three months (control period), followed by LCHF dietary intervention for the next three months (intervention period), or vice versa.

DETAILED DESCRIPTION:
Mitochondrial disease (MD) is a clinically and genetically heterogenous group of disorders. The dysfunction of the mitochondrial respiratory chain results in ATP shortage and energy depletion resulting in multi system disease. Therapeutic interventions are currently limited and focus on relieving symptoms, since no curative therapies exist. The m.3243A>G related MD is presumably the most frequent MD affecting at least 1 in 5000 people, and the MIDD (Mitochondrial Inherited Diabetes and Deafness) phenotype is its most frequent clinical phenotype. The role of nutrition, providing the essential nutrients for mitochondria to produce energy, is an important disease modifier in MIDD.

A ketogenic diet (KD) is a very low-carbohydrate ( ±20 grams a day) high-fat diet that shifts metabolism towards β-oxidation and ketone body production. In cell studies and mice models for MD, ketone bodies or KD significantly affect different dimensions of mitochondrial function. KD has been proven to effectively treat intractable epilepsy in children with MD. The investigators recently performed a 12 week pilot study with KD in 20 adults with different types of mtDNA related MD. The KD improved glucose tolerance, yielded less migraine, and alleviated gastrointestinal symptoms. Despite these positive effects, it proved the KD is a difficult diet to follow and only 8/20 participants finished the 12 week KD intervention. The individuals with m.3243A>G related MD had the longest diet adherence. Because of the positive effects, over half of all participants switched to the more feasible and less restrictive low carbohydrate (± 50-100 gram/dag), high fat (LCHF) diet after completing the study. The positive effect of KD on the subtype of m.3243A>G related MD was very recently confirmed in another study. The LCHF diet however provides no ketone bodies and its effect in mitochondrial disease is not studied properly yet.

In irritable bowel syndrome, specific dietary regimens as low-fermentable, oligo-, di-, monosaccharides and polyols (FODMAPs) but also LCHF diets are considered therapeutic. A diet low in fermentable carbohydrates reduces the fermentation by the gut microbiota and is therefore thought to reduce bloating and other gastro intestinal complaints. Based on the results of a previous study from the investigators and the effect of LCHF diets in irritable bowel syndrome, the investigators hypothesize the same positive effect in the cohort of m.3243A>G related MD in which gastro intestinal complaints are very common.

An adult diabetes team studied the gut microbiome and observed significant differences in various species and pathways between the faecal stool samples of diabetes patients and healthy controls, and that gut microbiome composition is associated with glycemic control. The gut microbiome is a very promising study field. More insight in patients gut microbiome and the way it can be altered with nutrition could lead to new treatment options and symptom relieve which is very relevant to MD patients. Therefore it is interesting to compare the gut microbiome of MIDD patients with already analysed stool samples of healthy controls and diabetes patients, and study the effect of an LCHF diet intervention.

The LCHF diet is an established treatment option in diabetes, with positive effects on glucose homeostasis. The investigators have initially chosen the subgroup of m.3243A>G related MIDD patients as they hypothesize that the LCHF could help slow down the progression of diabetes severity and reduce the necessity for treatment with insulin in these patients in particular. Since the team could not find enough participants with MIDD they intent to include also participants with MD caused by the m3243A>G mutation but without diabetes. These patients still have a lot of gastro intestinal problems as well as fatigue and headaches, all relevant symptoms that possibly can be affected with the low carbohydrate diet. So the primary outcomes as mentions in the title of the study: effect on clinical symptoms and the gut microbiome are relevant for this patient population aswell.

Studies in the heterogeneous patient population with MD are challenging. By choosing a relatively frequent genotype the investigators can minimize this problem and study a defined cohort. Additionally the investigators will use a cross over design ("patients being their own controls") to further decrease the number of patients needed to be included to achieve robust data.

Previous experience with trials in MD including patient consultations has led to an insight that the Goal Attainment Scaling (GAS) is an important individually tailored outcome for this patient group. With the GAS patients choose and score personal goals that they want to achieve with the diet intervention.

Taken together, The investigators intend to perform a pilot study to investigate the effect on clinical symptoms, as measured by GAS, as well as assessing gastrointestinal complaints and the impact on the gut microbiome of a low carbohydrate, high fat diet intervention. This study will focus on a cohort comprising adult patients exhibiting m.3234A>G mutation-related MD. Additionally, within the subgroup of patients with m.3234A>G-related MIDD, diabetes control will be also be evaluated.

1.1 Visits:

Visit baseline:

* Signing informed consent
* Final check inclusion and exclusion criteria
* Randomisation
* Secure baseline stool sample
* Check baseline food diary
* Vitals including blood pressure
* NMDAS , SF 12,
* GAS (Goal Attainment Scaling)
* Nutritional assessment: Weight, body composition (Multi frequency BIA SECA BCM 555)
* Online Questionnaires will be filled in Castor database during the visit under supervision of the researcher to prevent missing data. Questionaires include: Gastro intestinal complaints, + SF 12, CIS fatigue, diet tolerance, adverse effects and medication
* Laboratory examinations (CK, HBA1c, lipid profile, kidney function, transaminases, lactate, ketone bodies, metabolomics)
* Patient instructions on home measurements and if randomised in the intervention group diet instructions including safety instructions.

Visit 12 weeks:

* NMDAS with SF 12
* Vitals including blood pressure
* GAS (Goal Attainment scaling)
* Nutritional assessment: Weight, body composition (Multi frequency BIA SECA BCM 555).
* Online Questionnaires will be filled in Castor during the visit under supervision of the researcher to prevent missing data.
* Laboratory examinations (CK, HBA1c, lipid profile, kidney function, transaminases, lactate, ketone bodies, metabolomics)
* Check on the home measurements and if randomised in the control group diet instructions and if randomised in the intervention group instructions how to stop the diet.

Visit 24 weeks:

* NMDAS with SF 12
* Vitals including blood pressure
* GAS (Goal Attainment scaling)
* Nutritional assessment: Weight, body composition (Multi frequency BIA SECA BCM 555).
* Online Questionnaires will be filled in Castor during the visit under supervision of the researcher to prevent missing data.
* Laboratory examinations (CK, HBA1c, lipid profile, kidney function, transaminases, lactate, ketone bodies, metabolomics)
* Check on the home measurements and diet instructions for after the study based on patients wishes.

1.2 Home measurements:

* Diet adherence will be checked with a digital food diary 3 of days including one weekend day. At baseline, 11 weeks and 23 weeks.
* Fecal sampling at baseline, 12 weeks and 24 weeks.
* Accelerometery: Activ8® has to be worn on the upper leg for 1 week at the time: At baseline, 11 weeks and 23 weeks.
* Weight measurement once a week.
* Headache diary: Headaches need to be registered during the whole study
* Glucose monitoring will be done with sensor derived glucometrics at the last 10 days of both the intervention and the control period. Two times (20 days) in total. Exclusively conducted for MIDD patients. In MIDD patients without continuous glucose monitoring in the usual care (this are the patients without intensive insulin therapy) the sensor will be blinded.

1.3 Instructions:

* Instructions on when and how to fill in the online eating report.
* Instructions on how to wear the actometer at screening.
* Diet instructions at the visits in the intervention period and during weekly telephone (or videocall) consultations during the first 4 weeks of the diet and thereafter at week 8. Diet instructions by a specialist dietitian. The diet instructions consist of a personalized diet plan and a patient brochure with links to recipes accompanied by verbal instructions. Diet and, if necessary medication, will be adjusted in the first few weeks based on glucose levels in blood, complaints, practical questions and weight developments. This will be done in the same manner as in regular patient care for adult diabetic patients who start with the LCHF diet. Difference between this protocol and this study is that in the protocol a diabetic nurse takes care of the medication changes and in this study Dr. Rick Meijer is responsible, or in his absence another internist experienced in the treatment of MIDD. Additional telephone or e-health consultations (mijnRadboud) can be planned as frequent as necessary depending on the questions of the patient. A specialised metabolic dietician is available 5 days a week. In the week after the participant has to switch back to usual care there is a telephone meeting planned to make sure the transition went safely and al information is clear for the participant.
* Instructions on how to collect a faecal stool sample
* Instructions for the blinded continuous glucose monitoring. Participant have to apply the sensor at home in week 11 and week 23. Exclusively for MIDD patients who don't have continuous glucose monitoring already.
* Safety instructions on how to prevent hypoglycemia and how to act in case of a hypoglycemic incident. These instructions will be personalized based on individual diabetes medication and blood glucose levels, the protocol is used as guideline for these personalized instruction. This protocol is usual care in diabetes patient care and based on the national guidelines. The instructions included medication changes. The safety instructions on how to adapt the diet to hypoglycaemic events are included in the diet brochure.

Investigational treatment: Low carbohydrate high fat diet Low carbohydrate (50-100 grams/day). The LCHF restricts a wide range of carbohydrate rich foods including sweets, sugar, grains, starchy vegetables, sweet legumes, fruit juices and sweetened dairy foods and replacing them with non-starchy vegetables, red fruits, meat, poultry, seafood, eggs, oil, nuts, and non sweetened high fat dairy foods such as cheese, butter, cream and Greek 10% fat yoghurt. Choosing cuts of meat higher in fat and fats, and the use of low carb alternatives like low carb bread is encouraged. This diet is automatically high in protein. We don't want the carbohydrate restriction to be stricter than 50 grams a day because we want a feasible diet without de adverse events that a ketogenic diet (very strict carbohydrate restriction of 20 grams a day) has. The low carbohydrate high fat diet is part of the national diabetes guidelines and is frequently prescribed in overweight diabetes type 2 patients with insulin resistance.

METHODS 2.1 Measurements

The questionnaires The Gastrointestinal complaints Questionnaire contains questions on gastrointestinal complaints (7 point Likert scale) form a validated Dutch gastro intestinal questionnaire. We used this questionnaire in studies with mitochondrial disease before. For severity we use a Numerical Rating Scales (NRS) stool frequency, Bristol stool chart and laxative use is being checked.

The general study questionnaire in the intervention phase there will be questions on feasibility and diet tolerance, adverse events and questions on diabetes medication doses (insulin use).

* Quality of life: SF-12 questionnaire The SF-12 Health Survey (see F1.SF-12-Dutch) is a shorter version of the SF-36 Health Survey that uses 12 questions to measure functional health and self-administered well-being. SF12 takes approximately three minutes to complete and it is a practical, reliable and valid measure of physical and mental health. It is useful in large population health surveys or for applications that combine a generic and disease-specific health survey. SF 12 is available in multiple languages, including Dutch. It covers the following eight health domains: 1) Physical functioning 2) Limitations in usual role activities because of physical health problems 3) Bodily pain 4) General health perceptions 5) Vitality (energy / fatigue) 6) Limitations in social activities because of physical or emotional problems 7) Limitations in usual role activities because of emotional problems and 8) General mental health. Two subscales are derived from the SF-12: the Physical Component Summary (PCS) and the Mental Component Summary (MCS). These summary scales based on the SF-12 correlate very highly with the SF-36 version. The SF-12 uses norm-based scoring, so comparisons can be made among the other generic health surveys. The SF-12 and SF 36 are frequently used in mitochondrial disorders and it is advised to always combine the NMDAS with one of these quality of life questionnaires.
* Fatigue questionnaire: short checklist individual strength The Checklist Individual Strength is a 20-item self-reported questionnaire that captures four domains of fatigue: 1) subjective severity of fatigue 2) reduction in concentration, 3) reduction in motivation and 4) reduction in activity. Respondents will rate the extent to which each statement is true for them in the past two weeks on a seven-point Likert scale. The scores are summed up accordingly. The higher the score, the higher the fatigue level. A score between 27 and 35 suggests an increased risk for fatigue and a score above 35 suggests severe fatigue. The questionnaire has been used in various diseases, including mitochondrial diseases.

Questionnaires will be filled in digitally as eCRF in castor by the patients directly.

Nutritional Assessment: measurements will be performed according to our standard operation procedures Weight (kg), Weight loss (%), Height(cm) BMI (kg/m2) and body composition will be measured with bioimpedance analysis SECA BCM 555®. With the outcome variables: Fat percentage. Fat free Mass (FFM) (kg) and FFM Index (kg/m2), Skeletal muscle mass index (kg/m2) and phase angle(◦).

Blood test:

* creatinine kinase (CK),
* diabetes: HbA1c and home glucose monitoring (exclusively in MIDD patients)
* lipid profile (after overnight fast/or at least 4 hours of fasting): (triglycerides, high-density lipoprotein (HDL), low-density lipoprotein (LDL), total cholesterol),
* kidney function (MDRD), transaminases (ALAT and ASAT), lactate
* Ketones (beta-hydroxybutyric acid and acetoactetate)
* metabolomics

Home blood test:

Diabetes control assessments will be exclusively conducted for MIDD patients. Glucose monitoring can be done by blinded continues glucose monitors (Dexcom). Patients who are accustomed to glucose monitoring at home as part of their routine care will not be required to utilize the study-provided blinded monitor. Patients who use Insulin or glibenclamide, gliclazide, glimepiride or tolbutamine will be provided with a not blinded finger prick glucose meter to guarantee safety and to detect any low blood sugars in a timely manner. Measuring blood glucose with this home device with a finger prick is requested when participants experience complaints that may indicate low blood sugar, such as extreme hunger, sweating, trembling, dizziness, palpitations, yawning, being confused or feeling restless.

Three-day food record:

A digitally three-day food record is a self-reported account of all foods and beverages consumed by a respondent over three days, two working days and one day of the weekend. The data will be entered by the participant in the Eetmeter app.

The aim of the use of the food record is to finetune the diet and evaluate diet adherence. It helps patients to get more insight in their carbohydrate intake and to better manage the diet so they are free to use it more frequently (but for the study only 3 times 3 days are required). Intake will be automatically calculated in the eetmeter app. Data on energy (kcal), carbohydrates (gram), protein (gram) fat (gram), fibre (grams) and water (ml) intake will be registered.

Accelerometry:

The Activ8 is used to measure average metabolic equivalents(METS) over one week period. Activ8 and the elaborate use instructions will be sent to patients' home (see E4.Draaginstructie Activ8 actometer). Patients will apply the actometer and wear activ8 for one week during 24 hours per day. The device waterproof so the participants can also wear it during shower or swimming. Actometer activ8 has to be worn on the upper leg for 1 week at the time in total 3 times: during the screening, week 6, and week 12. This is used to calculate the energy expenditure for the individual diet advice[29] since the amount of activity can be a confounder as well as an possible efficacy variable. Actometry is considered the gold standard for activity measurements and it is a non-invasive method[30].

NMDAS:

The Newcastle Mitochondrial Disease Scale for Adults (NMDAS) is a semi-quantitative clinical rating scale designed specifically for all forms of mitochondrial disease. It was developed and tested in Newcastle with the aim of providing a validated and reproducible measurement of disease progression. It is now the most widely used outcome measure in clinical trials for mitochondrial disease. The NMDAS scale considers many parameters, including neurological disease, diabetes, cardiac involvement. The NMDAS need to be filled during the screening and week 12 by the metabolic specialist directly in castor.

Headache diary Frequency and severity of headages are scored with a headaches diary. Headaches need to be registered only if occur. A NBS score for severity of the headache and if patients took medication for the headache can be registered in the diary.

Other study parameters:

Patient characteristics: age, gender.

2.2 Randomisation, blinding and treatment allocation After signing informed consent participants will be randomized in the intervention or control group with the castor database. There is no blinding or treatment allocation in this study. Upon arrival on the screening, the participants receive an ID code. The first participant will be number one and so on.

2.3 Withdrawal of individual subjects Subjects can leave the study at any time for any reason if they wish to do so, without affecting future management and treatment. The investigator can decide to withdraw a subject from the study for urgent medical reasons.

2.4 Replacement of individual subjects after withdrawal Patients will not be replaced after withdrawal. However, if patients do not meet the inclusion and exclusion criteria based on the results from the first visit, then these patients will be replaced.

2.5 Follow-up of subjects withdrawn from treatment Patients will be asked if they are willing to complete the final study visit after they stopped the diet. They are asked why they stopped the diet but they are not obligated to answer this or come to the closing visit.

3. STATISTICAL ANALYSIS

Descriptive analyses Statistical analysis will be performed using SPSS statistics version 24 (IBM). Baseline characteristics will be reported, at timepoint 0 weeks, as means ± SD for normally distributed variables, as median and IQR for non-normally distributed variables and as a percentage of the total population for the categorical variables.

ELIGIBILITY:
Inclusion Criteria:

* Mitochondrial disease caused by the m.3243A>G mutation m.3243A>G mutation
* BMI ≥ 18.5 kg/m2
* Good cognitive health

Exclusion Criteria:

* Kidney failure (MDRD <60 or proteinuria)
* Use of SGLT2-inhibitors
* Already on a carbohydrate restricted diet at baseline (carbohydrate intake <100 grams per day)
* Pregnancy

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 17 (Actual)
Dates: Start 2024-01-05 (Actual); Primary Completion 2025-01-03 (Actual); Study Completion 2025-01-03 (Actual)

PRIMARY OUTCOMES:
Goal Attainment Scaling (GAS) | 12 weeks
  The Goal Attainment Scale (GAS) is an individualized outcome measure involving goal selection and goal scaling that is standardized in order to calculated the extent to which a patient's goals are met. The scores can range from -2 to +2 with 1-point increments. A score of 0 indicates that the expected level is reached. A negative score means that the level reached was lower than expected, and can be classified as lower (-1) of much lower (-2). A positive score means that the level reached was higher than expected, and can be classified as higher (+1) of much higher (+2).
Faecal microbiome composition analyses via DNA isolation | 12 weeks
  The faecal microbiome composition of the participants with their usual diet will be compared the faecal microbiome composition after adhering to the low-carbohydrate high-fat diet. More specifically, DNA will be isolated from the stool samples, and will be compared between the intervention period and the control period.

SECONDARY OUTCOMES:
Glucose monitoring | 12 weeks (home glucose monitoring for two time periods of 10 days)
  Glucose monitoring will be performed with a glucose monitoring device that a participant will wear for two time periods of 10 days. One time period will be at the end of the intervention period, and one time period at the end of the control period. The time in range, periods of hypoglycemia and periods of hyperglycemia will be determined. This will exclusively conducted for MIDD patients. In MIDD patients without continuous glucose monitoring in the usual care (this are the patients without intensive insulin therapy) the sensor will be blinded.
Gastrointestinal complaints questionnaire | 12 weeks
  Questionnaire including a numerical score on severity of gastrointestinal complaints (1 = not severe and 10 = very severe), stool frequency, stool type determined via the Bristol stool chart and laxative use.
Diet adherence | 3 days
  Digital food diary of three days, including one weekend day
Checklist Individual Strength (CIS) | 12 weeks
  The Checklist Individual Strength is a 20-item self-reported questionnaire that captures four domains of fatigue: 1) subjective severity of fatigue 2) reduction in concentration, 3) reduction in motivation and 4) reduction in activity. Respondents will rate the extent to which each statement is true for them in the past two weeks on a seven-point Likert scale. The scores are summed up accordingly. The higher the score, the higher the fatigue level. A score between 27 and 35 suggests an increased risk for fatigue and a score above 35 suggests severe fatigue.
Newcastle Mitochondrial Disease Adult Scale (NMDAS) | 12 weeks
  The NMDAS has been introduced to allow evaluation of the progression of mitochondrial disease in adult patients over 16 years. The rating scale encompasses all aspects of mitochondrial disease by exploring several domains: Current Function; System Specific Involvement; Current Clinical Assessment and Quality of Life.
  Each question in the NMDAS has a possible score from 0-5. Each of the first 3 domain scores are calculated by simply summing the scores obtained for each question in that section. The higher the score the more severe the disease. The Quality of Life will be assessed with the Short Form (SF)-12. The SF-12 is a self-reported outcome measure assessing the impact of health on an individual's everyday life.
Accelerometry | 7 days
  Physical activity measurement to calculate the Physical Activity Level (PAL)
Headache diary | 12 weeks
  Reporting frequency of headaches and use of medication for headaches
Bodyweight measurements | 1 week
  Bodyweight of participants will be measured
Body Mass Index (BMI) | 12 weeks
  Body Mass Index (BMI) will be determined during every visit
Bio-electrical Impedance Analysis (BIA) | 12 weeks
  Body composition will be measured with bioimpedance analysis, with the goal to determine body muscle mass and body fat mass.
Creatine Kinase (CK) | 12 weeks
  Creatine Kinase levels in the blood will be measured (physiological parameter)
Hemoglobin A1c (HbA1c) | 12 weeks
  Hemoglobin A1c (HbA1c) levels in the blood will be measured (physiological parameter)
Lipid profile blood test | 12 weeks
  The lipid profile in the blood will be determined after at least 4 hours of fasting. The lipid profile includes triglycerides, high-density lipoprotein (HDL), low-density lipoprotein (LDL) and total cholesterol (physiological parameters)
Liver function blood test | 12 weeks
  The transaminase levels in the blood will be determined to assess liver function. These include the alanine aminotransferase (ALAT) and Aspartate transaminase (ASAT) values (physiological parameters)
Kidney function blood test | 12 weeks
  Creatinine levels in the blood will be determined (physiological parameter), which will be used to calculate the Modification of Diet in Renal Disease (MDRD). The MDRD is a measure for glomerular filtration rate (GFR) based on creatinine and patient characteristics.
Blood lactate concentration | 12 weeks
  Lactate levels in the blood will be determined (physiological parameter)
Blood ketone concentration | 12 weeks
  Ketone levels (specifically beta-hydroxybutyrate) in the blood will be determined with a finger prick (physiological parameter)

CONTACTS AND LOCATIONS:
Overall Officials: Heidi Zweers- van Essen, Doctor, Principal Investigator — Radboud University Medical Center
Locations (1):
- Radboudumc, Nijmegen, Gelderland, Netherlands

IPD SHARING:
Plan to Share IPD: No